CLINICAL TRIAL: NCT05189028
Title: Phase III Randomized Prospective Clinical Study of Neoadjuvant Chemotherapy With Gemcitabine and Cisplatin(GP) Versus Definite Cisplatin Combined Weekly Chemoradiotherapy for Locally Advanced Bulk Cervical Cancer
Brief Title: Study of Neoadjuvant Chemotherapy Versus Definite Concurrent Chemoradiotherapy for Locally Advanced Bulk Cervical Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chuangzhen Chen (Other)
Responsible Party: Sponsor-Investigator, Chuangzhen Chen, Deputy Director, Department of Radiation Oncology, Shantou University Medical College
Organization: Shantou University Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NACT-CC-001
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Cervical Cancer; Neoadjuvant Chemotherapy
Keywords: Cervical Cancer; NACT(Neoadjuvant Chemotherapy); Locally Advanced Bulk Cervical Cancer; Chemoradiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Locally advanced bulk cervical cancer neoadjuvant chemotherapy group(NACT) (Experimental): Radiation: Radiotherapy with IMRT/VMAT+192Ir-HDR brachytherapy Radiotherapy: 46Gy/23F to external pelvic radiotherapy and 14Gy/7F boost to imaging diagnosis of positive lymph nodes 192Ir-HDR brachytherapy:A Point dose 6Gy*4-6F
  Drug: gemcitabine plus cisplatin,cisplatin Neoadjuvant chemotherapy:gemcitabine and cisplatin (GP) regimen*2 cycles Concurrent Chemotherapy: Weekly cisplatin chemotherapy ≥5 cycles
  Interventions: Drug: gemcitabine and cisplatin
- Locally advanced bulk cervical cancer chemoradiotherapy group(CCRT) (Active Comparator): Radiation: Radiotherapy with IMRT/VMAT+192Ir-HDR brachytherapy Radiotherapy: 46Gy/23F to external pelvic radiotherapy and 14Gy/7F boost to imaging diagnosis of positive lymph nodes 192Ir-HDR brachytherapy:APoint A dose 6Gy*4-6F
  Drug: cisplatin Concurrent Chemotherapy: Weekly cisplatin chemotherapy ≥5 cycles
  Interventions: Drug: gemcitabine and cisplatin

INTERVENTIONS:
Drug: gemcitabine and cisplatin — Neoadjuvant chemotherapy:gemcitabine and cisplatin

SUMMARY:
This phase III randomized prospective clinical study was conducted to compare the short-term and long-term outcomes of gemcitabine and cisplatin neoadjuvant chemotherapy versus definite cisplatin weekly concurrent chemoradiotherapy in patients with locally advanced bulk cervical cancer.

DETAILED DESCRIPTION:
Platinum-based concurrent chemoradiotherapy is the standard of care recommended by the NCCN for locally advanced cervical cancer of stage IB3, IIA2 and IIB-IVA (2018 FIGO stage) (cervical tumor ≥4cm). The 5-year survival rate of concurrent chemoradiotherapy for locally advanced cervical cancer has been reported in foreign literatures at 64.5-67%. The 3 - and 5-year survival rates of the concurrent chemoradiotherapy in our hospital were 78.6% and 70.5%, respectively, while the 3 - and 5-year survival rates of the concurrent chemoradiotherapy with cisplatin monotherapy were 66.4% and 63.1%, respectively. In the concurrent radiotherapy and chemotherapy, although many studies have tried paclitaxel, irinotecan, gemcitabine and other concurrent radiotherapy and chemotherapy with cisplatin, some encouraging results have been obtained, but at the same time, more obvious toxic and side effects have also appeared in the combination drug. At present, there is no evidence that the combined use of these radiotherapy sensitizers is superior to the single use of cisplatin. Adjuvant chemotherapy also did not show a survival advantage.

Neoadjuvant chemotherapy (NACT) is a systemic chemotherapy given before local treatment of malignant tumors (surgery or radiotherapy), mainly used for the treatment of breast cancer, cervical cancer, and solid head and neck tumors. Neoadjuvant chemotherapy plus surgery in locally advanced cervical cancer research more, but there is no specification of neoadjuvant chemotherapy plus radiation and chemotherapy research reports. Possible benefits of neoadjuvant chemotherapy: 1. Reduce tumor volume, reduce tumor displacement during radiation, and thus reduce the radiation dose to surrounding normal tissues (rectum, bladder, etc.); 2. Reduce the proportion of hypoxic cells and increase the radiotherapy sensitivity; 3. Suppression or elimination of micrometastatic lesions may exist in the whole body, and can prevent distant metastasis.

Rydzewska et al. conducted a large sample study showing that neoadjuvant chemotherapy can prolong overall survival and progression-free survival. For early and locally advanced cervical cancer, neoadjuvant chemotherapy combined with radical surgery is more meaningful than surgery alone. He et al. reported on 62 cases of Ⅰ b2 ~ Ⅱ b stage cervical cancer patients with paclitaxel plus cisplatin 2-3 courses of neoadjuvant chemotherapy, the total effective rate was 90.32%, among them the complete response rate was 30.65%, tumor after chemotherapy significantly smaller.

Gemcitabine (GEM) is a synthetic nucleoside derivative of cytosine, which mainly acts on S phase and has been used in solid tumors for more than 20 years. Duenas-Gonzalez et al. reported that gemcitabine combined with cisplatin induced chemotherapy in the primary treatment of locally advanced (IB2-IIIB) cervical cancer stage II study, the total response rate of induction chemotherapy plus surgery was 95% (7.5%CR and 87.5%PR), grade 3-4 granulocytopenia accounted for 13.8% and 3.4%, and non-hematological toxicity was slight. Therefore, the chemotherapy response rate of GP(gemcitabine/cisplatin) regimen was similar to that of PC (paclitaxel/cisplatin) regimen in cervical cancer, but the side effects were relatively small.

IMRT/VMAT modern precision radiotherapy technology is more and more popular in the radiotherapy of cervical cancer, precision radiotherapy has better conformal, can significantly reduce the external radiation dose of pelvis and small intestine; It is also possible to reduce the dose and volume of surrounding normal tissues (rectum, bladder, etc.) during target mapping and planning. However, the local tumor of the massive cervical cancer is huge, and the volume of the surrounding normal tissue decreases significantly during the radiotherapy and chemotherapy during irradiation, which results in increased displacement change of the surrounding normal tissue, so that the normal tissue outside the target area during the planning and design enters the irradiation field, and weakens the benefits of precise radiotherapy technology. Neoadjuvant chemotherapy reduces local cervical tumors in advance, improves tumor hypoxia and reduces tumor displacement during concurrent chemoradiotherapy. Theoretically, it has obvious benefits to reduce side effects in normal tissues around the week.

This study attempted to administer gemcitabine and cisplatin (GP) regimen neoadjuvant chemotherapy in large locally advanced cervical cancer, with the expectation that the neoadjuvant chemotherapy group could improve the local control rate, reduce the distant metastasis rate, and reduce the side effects of radiotherapy in normal tissues, thus improving the overall survival rate, and providing a scientific basis for the development of a rational, effective, low-toxicity, individualized comprehensive treatment plan suitable for modern precise radiotherapy technology for locally advanced cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of primary cervical squamous cell carcinoma, adenocarcinoma, or adenosquamous cell carcinoma.
* According to the 2018 International Federation of Cervical Cancer Obstetrics and Gynecology (FIGO) staging standard, the patient was diagnosed with local tumor ≥4cm in stage IB3, IIA2, IIB-IVA by at least one expert with associate high degree or above in the department of gynecology and gynecology.
* Age≥18 & ≤70.
* ECOG score 0-2.
* WBC ≥4.0×109/L, hemoglobin ≥60g/L, platelet ≥100.0×109/L; Serum bilirubin ≤ upper limit of normal, ALT, AST, ALP ≤ upper limit of normal ×2.5; Urea nitrogen (BUN) ≤ upper limit of normal ×1.5, creatinine (Cr)≤ upper limit of normal ×1.5.
* Patients with prior malignancy are eligible if disease-free ≥ 5 years.
* Signed study-specific informed consent form prior to study entry.

Exclusion Criteria:

* Line has anti-tumor treatment, including chemotherapy, radiotherapy, surgery).
* Stage Ia1- IB2 and IVB cervical cancer.
* Patients with uncontrolled serious medical or mental illnesses.
* Women in pregnancy or lactation.
* Psychological, family, social factors, such as lead to no informed consent.
* Into the group of the first five years in addition to the cervical cancer merger other patients with a history of malignant tumor.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years

SECONDARY OUTCOMES:
Local-regional control | 2 years
Distant metastasis-free survival | 2 years
Disease-free survival | 2 years after randomization
Acute and late toxicities using CTCAE v4.0 | 2 years
  The probabilities of grade ≥ 3 acute toxicities and 2-year late toxicities of bladder and rectum.

CONTACTS AND LOCATIONS:
Overall Officials: Chuangzhen Chen, MD, Principal Investigator — Cancer Hospital, Shantou University Medical College
Locations (1):
- Cancer Hospital, Shantou University Medical College, Shantou, Guangdong, China